CLINICAL TRIAL: NCT04363658
Title: Efficacy Study of Shunt Operation in Patients With Disorder of Consciousness of Post-traumatic Hydrocephalus (PTH) by Methods of Neuroelectrophysiology
Brief Title: Efficacy Study of Hydrocephalus Surgery by Methods of Neuroelectrophysiology
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: 202001015
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Hydrocephalus
Keywords: neuroelectrophysiology; hydrocephalus; disorder of consciousness
MeSH Terms: conditions — Hydrocephalus; Consciousness Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The symptoms of hydrocephalus containing consciousness condition with muscle tone in some patients will be relieved, after the cerebrospinal fluid release test is carried out. Neuroelectrophysiology in patients with disorders of consciousness of post-traumatic hydrocephalus (PTH) can establish the association with consciousness and muscle tone to a certain extent, and predict the shunt effect of PTH with disorders of consciousness.

ELIGIBILITY:
Inclusion Criteria:

Patients with disorder of consciousness in traumatic brain injury. The presence of hydrocephalus through image examination.

Exclusion Criteria:

Patients who cannot tolerate shunt surgery. Sedation maintained by greater than 0.15mg/kg/hour of midazolam or the infusion dose of propofol higher than 4mg/kg/hour.

Patients who are participating in drug research or other clinical trials.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient age from 16 to 70 years
Sampling Method: Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2020-05-10 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Score of glasgow outcome scale in 6 months after shunt operation | 6 months

SECONDARY OUTCOMES:
Score of glasgow outcome scale in 6 months after shunting under different ventricular pressure | 6 months
Revised coma recovery scale (CRS-R) in 1 week after shunting | 1 week
Modified Ashworth Scale (MAS) in 1 week after shunting | 1 week
Revised coma recovery scale (CRS-R) in 1 month after shunting | 1 month
Modified Ashworth Scale (MAS) in 1 month after shunting | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Nicolet EEG, Pleasanton, California, United States